CLINICAL TRIAL: NCT05307107
Title: Recognize the Power Within and SHINE - Educators' Digital Occupational Well-being Intervention in Health and Social Care Education
Brief Title: Educators' Digital Occupational Well-being Intervention During Working Hours
Acronym: SHINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: The Trade Union of Education in Finland (OAJ) (Unknown); University of Eastern Finland (Other)
Responsible Party: Principal Investigator, helena Leino-Kilpi, Professor, University of Turku
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: University of Turku_UTurku
Record Dates: First submitted 2022-01-12; First posted 2022-04-01 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Well-being; Physical Activity; Recovery; Self Regulation
Keywords: educator; occupational well-being; working hours; physical activity; intervention; recovery; break
MeSH Terms: conditions — Motor Activity; Self-Control

STUDY DESIGN:
Intervention Model Description: Participants (n=80) are educators working in health and social care education in secondary level education in five different educational organizations, which have similar management systems and providing time-support to implement SHINE during working hours. Organizations are randomly assigned either in intervention group (IG, n=2) receiving SHINE or in control group (CG, n=3) without the program continuing their normal daily routines receiving SHINE for their voluntary use after this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (IG) (Experimental): Participants are educators working in health and social care education receiving 8 work week-SHINE.
  Interventions: Behavioral: SHINE
- Control group (CG) (No Intervention): Participants are educators working in health and social care education without the program continuing their normal daily routines receiving SHINE for their voluntary use after this study (waitlist).

INTERVENTIONS:
Behavioral: SHINE — Intervention group will use a 8-workweeks the digital Smart Break SHINE program with workplace support (encouragement and time-support) including daily 3 minutes break exercises twice a day; 1) physical exercise - break and 2) body/mind breathing exercise - break earning stars for exercise completed. The program includes weekly self-reflective task of individual well-being during working hours with weekly changing theme (avoiding sitting time, nature benefits, relaxation exercises, increasing physical activity in workplace etc.) earning diamonds for every weekly task completed. Participants self-monitors their weekly individual resources levels asked in every Thursday (1-5, 1= very poor. 5= very good). Program includes e-mail remainders set by participant themselves for suitable time frame These individual well-being actions takes approximately 15 minutes/workday. Control group will receive this program after this study (waitlist protocol).
  Arms: Intervention group (IG)

SUMMARY:
This controlled quasi experimental intervention study follows the MRC framework for complex interventions (Bleijenberg et al. 2018) aiming to promote educators' individual aspect of occupational well-being. The purpose of this study is: 1) to evaluate the effectiveness of 8-workweek SHINE (= Self-Help INtervention for Educators) on educator's individual aspect of occupational well-being comparing intervention and control groups and 2) to describe the possible associating factors for the effectiveness of the intervention (if any) and 3) to evaluate SHINE's acceptability (utility and usability) within intervention group.

DETAILED DESCRIPTION:
Overall Occupation Well-being (OW) is seen through four aspects of working life: 1) workers's resources and work (individual aspect), 2) work community, 3) working conditions and 4) professional competence (Saaranen et. al 2007). This study focuses in the individual aspect of OW, worker's resources and work and associating factors. This evidence base digital SHINE intervention is conducted in Finland within five different social and health care educational organizations randomly allocated either in intervention group (n=2) or in control group (n=3). Participants are working as qualified full-time educators in these organizations; intervention group (n=39) and control group (n=41). The intervention consists of four components: 1) physical activity, 2) recovery, 3) self-regulation and 4) workplace support designed to promote worker's resources at work. First three of these components are in digital program called, Smart Break SHINE. Educators' does short 3 minute exercises twice/workday (movement and breathing mind/body exercises) and additionally completes weekly reflective wellness actions during working hours. Last component, workplace support, comes from educators' organizations enabling time support and encouraging educators' to conduct these exercises during working hours taking approximately 10-15 min/workday. Control group continues their normal daily routines without this program.

Aim of this intervention is to promote educators' individual aspect of occupational well-being, the balance between individual resources and workload factors, during working hours. Main outcome is resource-workload-balance (RSW) and heart rate variability (HRV) and secondary outcomes are general well-being (GW) and overall occupational well-being (OW). Other outcomes are SHINE-components being associating factors in individual aspect of OW, physical activity, recovery, self-regulation and workplace support (condition outcomes). Also the usability and utility of the intervention is studied from the intervention group after using the program 8 workweeks.

ELIGIBILITY:
Inclusion Criteria:

* Working as qualified educator (at least qualification of EQF 7) in secondary health and social care education
* Full-time work contract
* Having at least one-year employment in the organization

Exclusion Criteria:

* having pacemaker or being pregnant (cause of the HRV measures)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-05-29 (Actual)

PRIMARY OUTCOMES:
Change in resource-workload-balance | pre (week before enrollment) /post (after 8-workweeks) /follow-up (after 12 weeks of enrollment)
  Change in resource-workload-balance. 16-item self-reported questionnaire with continuous scale 1-5 (1= very poor - 5= very good).
  Questionnaire consists of questions of personal resources at work and workload factors [9-item developed for this study and 7 items from "Occupational well-being of social and health care teachers - index questionnaire" (Saaranen et al., 2007)]
Change in HRV | pre (week before enrollment) /post (after 8-workweeks) /follow-up (after 12 weeks)
  Change in physical heart rate variability (=HRV). Change in the HRV (try to increase heart rate variability); in the variation in the time interval between consecutive heartbeats in milliseconds (ms).
  Heart rate variability (HRV) 3 minutes measurements are performed in work mornings at rest using Kubios HRV mobile application and a compatible belt-heart rate sensor (Polar H10 or H7). The beat-to-beat RR interval data (i.e. time intervals between successive heart beats) is pre-processed and analyzed at Kubios (Tarvainen et al. 2014; https://www.kubios.com/)

SECONDARY OUTCOMES:
Change in Overall occupational well-being | pre (week before enrollment) /post (after 8-workweeks) /follow-up (after 12 workweeks)
  Change in overall occupational well-being With one item: " I feel that my personal occupational well-being in this profession compared to the best possible level is" (continuous scale 0-5, 0= very poor - 5 = very good) from 'Occupational well-being of social and health care teachers - index questionnaire' (Saaranen et al., 2007).
Change in General well-being | pre (week before enrollment) /post (after 8 workweeks) /follow-up (after 12 workweeks)
  Change in individual's well-being in general. With 5-item "WHO5 well-being index-questionnaire" (https://www.corc.uk.net/outcome-experience-measures/the-world-health-organisation-five-well-being-index-who-5/).
  The WHO-5 consists of five statements, which respondents' rate according to the scale 0-5 (in relation to the past two weeks, 0= at no time- 5= all the time). The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.

OTHER OUTCOMES:
Change of Physical activity_condition | pre (week before enrollment) /post (after 8-workweeks) /follow-up (after 12 workweeks)
  Change of physical activity during working hours (etc. less sitting). Intervention's component with 3-item "OSPAQ, occupational sitting and physical activity questionnaire" (CHAU et al., 2012) including questions of weekly working hours (h) and working days (d) and physical activity at work with percentages during that week (100 % is total activity in workweek consisting, sitting, standing, walking and heavy labour).
Change of Recovery_condition | pre (week before enrollment) /post (after 8-workweeks) /follow-up (after 12 workweeks)
  Intervention's component: 4-item recovery measurement (psychological detachment and relaxation) adapted from "Recovery experience questionnaire" (Sonnentag & Fritz, 2007). Likert scale 1-5 (1= total disagreement to 5= total agreement, 5 indicating better recovery). Recovery measured during working hours (de Bloom et al. 2015).
Change of Self-regulation_condition | pre (week before enrollment) /post (after 8-workweeks) /follow-up (after 12 workweeks)
  Intervention's component:
  6-item developed for this study based on previous references (etc. Hennessy et al., 2020) with continuous scale 1-5 (1= total disagreement to 5= total agreement, 5 indicating better self-regulation of personal resources at work)
Change of Workplace support_condition | pre (week before enrollment) /post (after 8-workweeks) /follow-up (after 12 workweeks)
  Intervention's component: 2-item developed for this study from the previous studies indicating the importance providing support towards personal resources during working hours (etc. Arian et al., 2018 and Singh et al., 2019). Continuous scale 1-5 (1= total disagreement to 5= total agreement, 5 indicating better support towards personal resources).
Background variables | pre (week before enrollment)
  Background variables:
  5-item personal related (age, gender and family relations) 5-item work-related (work experience, remote working and work autonomy and vacations during intervention time)
SHINE Acceptability: usability (intervention group) | post 8-workweeks
  With 10-item SUS-scale (system usability scale) (Brooke, 1996) of the Smart Break SHINE program's usability. Likert scale 1-5 (1= strongly disagree- 5= strongly agree).There is specific formula to o calculate to obtain the overall value of SUS range of 0 to 100, 100 being the best SUS score for occupational well-being program, Smart Break-SHINE.
SHINE Acceptability: usefulness (intervention group) | post 8-workweeks
  9-item The utility and actions for development of SHINE developed for this study is based on Medical Research Council (MRC) guidance for the process evaluation of complex interventions (Moore et al., 2015).
  Continuous scale 1-5 (1= strongly disagree- 5= strongly agree, 5 indicating better usefulness of the program) and two open-ended questions with no subjective opinions of the best qualities of SHINE and actions for development.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Leino-Kilpi, PhD, Study Director — University of Turku
Locations (1):
- Jenni Rinne, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
This data is available only for this study

REFERENCES:
- [Background] Bleijenberg N, de Man-van Ginkel JM, Trappenburg JCA, Ettema RGA, Sino CG, Heim N, Hafsteindottir TB, Richards DA, Schuurmans MJ. Increasing value and reducing waste by optimizing the development of complex interventions: Enriching the development phase of the Medical Research Council (MRC) Framework. Int J Nurs Stud. 2018 Mar;79:86-93. doi: 10.1016/j.ijnurstu.2017.12.001. Epub 2017 Dec 5. PMID 29220738
- [Background] Tarvainen MP, Niskanen JP, Lipponen JA, Ranta-Aho PO, Karjalainen PA. Kubios HRV--heart rate variability analysis software. Comput Methods Programs Biomed. 2014;113(1):210-20. doi: 10.1016/j.cmpb.2013.07.024. Epub 2013 Aug 6. PMID 24054542
- [Background] Sonnentag S, Fritz C. The Recovery Experience Questionnaire: development and validation of a measure for assessing recuperation and unwinding from work. J Occup Health Psychol. 2007 Jul;12(3):204-21. doi: 10.1037/1076-8998.12.3.204. PMID 17638488
- [Background] Chau JY, Van Der Ploeg HP, Dunn S, Kurko J, Bauman AE. Validity of the occupational sitting and physical activity questionnaire. Med Sci Sports Exerc. 2012 Jan;44(1):118-25. doi: 10.1249/MSS.0b013e3182251060. PMID 21659903
- [Background] de Bloom J, Kinnunen U, Korpela K. Recovery Processes During and After Work: Associations With Health, Work Engagement, and Job Performance. J Occup Environ Med. 2015 Jul;57(7):732-42. doi: 10.1097/JOM.0000000000000475. PMID 26147541
- [Background] Hennessy EA, Johnson BT, Acabchuk RL, McCloskey K, Stewart-James J. Self-regulation mechanisms in health behavior change: a systematic meta-review of meta-analyses, 2006-2017. Health Psychol Rev. 2020 Mar;14(1):6-42. doi: 10.1080/17437199.2019.1679654. PMID 31662031
- [Background] Arian M, Soleimani M, Oghazian MB. Job satisfaction and the factors affecting satisfaction in nurse educators: A systematic review. J Prof Nurs. 2018 Sep-Oct;34(5):389-399. doi: 10.1016/j.profnurs.2018.07.004. Epub 2018 Jul 7. PMID 30243696
- [Background] Singh C, Cross W, Munro I, Jackson D. Occupational stress facing nurse academics-A mixed-methods systematic review. J Clin Nurs. 2020 Mar;29(5-6):720-735. doi: 10.1111/jocn.15150. Epub 2020 Jan 2. PMID 31856356
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Background] Saaranen T, Tossavainen K, Turunen H, Kiviniemi V, Vertio H. Occupational well-being of school staff members: a structural equation model. Health Educ Res. 2007 Apr;22(2):248-60. doi: 10.1093/her/cyl073. Epub 2006 Jul 31. PMID 16880218
- See also: HRV measurement application — https://www.kubios.com/
- See also: WHO-5 scale: general well-being — https://www.corc.uk.net/outcome-experience-measures/the-world-health-organisation-five-well-being-index-who-5/
- See also: Brooke, 1996. SUS-scale: "Quick and dirty usability scale" — https://books.google.fi/books?hl=fi&lr=&id=IfUsRmzAqvEC&oi=fnd&pg=PA189&ots=GbmwBgnr1p&sig=F_eBa9DXsT6V_x9I8ZxhHsVgwG4&redir_esc=y#v=onepage&q&f=false